CLINICAL TRIAL: NCT01927198
Title: A Phase 2, Randomized, Double-Blind, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of RDEA3170 Monotherapy in Subjects With Gout
Brief Title: RDEA3170 Monotherapy in Subjects With Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDEA3170-201
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — verinurad

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- RDEA3170 5 mg qd (Experimental): No titration.
  Interventions: Drug: RDEA3170 5 mg
- RDEA3170 10 mg qd (Experimental): Increase from RDEA3170 5 mg to RDEA3170 10 mg qd at Week 2.
  Interventions: Drug: RDEA3170 10 mg
- RDEA3170 12.5 mg qd (Experimental): Increase from RDEA3170 10 mg to RDEA3170 12.5 mg qd at Week 4.
  Interventions: Drug: RDEA3170 12.5 mg
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: RDEA3170 5 mg
  Arms: RDEA3170 5 mg qd
Drug: RDEA3170 10 mg
  Arms: RDEA3170 10 mg qd
Drug: RDEA3170 12.5 mg
  Arms: RDEA3170 12.5 mg qd

SUMMARY:
This study will assess the serum uric acid lowering effects and safety of 3 dose levels of RDEA3170 compared to placebo in subjects with gout.

DETAILED DESCRIPTION:
This monotherapy study is the initial Phase 2 study for RDEA3170 and is designed to compare the safety and efficacy of multiple dose levels of RDEA3170 with placebo when given for up to 24 weeks to subjects with gout. The placebo control for RDEA3170 is included in this study to minimize bias in study assessments and monitoring. Further, to accomplish the goal of understanding the safety profile of RDEA3170, it is important to compare RDEA3170 monotherapy with placebo for at least 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets the diagnosis of gout per the American Rheumatism Association Criteria for the Classification of Acute Arthritis of Primary Gout.
* Subject has a serum urate level ≥ 6.5 mg/dL and ≤ 10.0 mg/dL during the Screening Period.
* Subject has a body mass index < 40 kg/m2.

Exclusion Criteria:

* Subject is pregnant or breastfeeding. Subject consumes more than 14 drinks of alcohol per week (eg, 1 drink = 5 oz [150 mL] of wine, 12 oz [360 mL] of beer, or 1.5 oz [45 mL] of hard liquor).
* Subject has a history or suspicion of kidney stones.
* Subject has a history or suspicion of drug abuse within the past 5 years.
* Subject has a history of symptomatic myositis/myopathy or rhabdomyolysis.
* Subject has a known or suspected human immunodeficiency virus infection.
* Subject has a positive test for active hepatitis B or hepatitis C infection.
* Subject has a history of malignancy within the previous 5 years with the exception of non-melanoma skin cancer that has been treated with no evidence of recurrence, treated cervical dysplasia, or treated in situ Grade 1 cervical cancer.
* Subject within the last 12 months with: unstable angina, New York Heart Association class III or IV heart failure, myocardial infarction, stroke, or deep venous thrombosis; or subjects currently receiving anticoagulants.
* Subject has a QT interval corrected for heart rate according to Fridericia's formula > 450 msec during the Screening Period, confirmed by a repeat assessment.
* Subject has uncontrolled hypertension.
* Subject has an estimated creatinine clearance < 60 mL/min.
* Subject has an alkaline phosphatase > 2.0 x upper limit of normal during the Screening Period.
* Subject has active liver disease or impaired hepatic function.
* Subject is receiving chronic treatment with more than 325 mg salicylates per day.
* Subject has a medical condition that requires or may require systemic immunosuppressive (eg, chronic low-dose oral prednisone) or immunomodulatory treatment.
* Subject is unable to take colchicine for gout flare prophylaxis.
* Subject is receiving strong or moderate CYP3A inhibitors, p-glycoprotein inhibitors, or digoxin.
* Subject received any strong enzyme- inducing drug or product (eg, rifampin, rifabutin, phenytoin, phenobarbital, St. John's Wort) within 2 months prior to Day 1 or refuses to refrain from taking these medications until the end of the study.
* Subject received an investigational therapy within 30 days or 5 half-lives (whichever is longer) prior to the Screening Period.
* Subject has any other medical or psychological condition, which in the opinion of the Investigator and/or Medical Monitor, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of RDEA3170 monotherapy at Week 12 | Week 12
  Percent change from baseline in serum urate levels at Week 12.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events and change from baseline in laboratory values, vital signs, and electrocardiograms | 8 months
  Safety assessments include adverse event (AE) recording, gout flare recording, clinical safety laboratory tests (eg, hematology, serum chemistry, and urinalysis), physical examinations, vital sign measurements, and ECGs.
Efficacy of RDEA3170 monotherapy at Week 24 | Week 24
  Percent change from baseline in serum urate levels at each visit. Proportion of subjects with a serum urate level < 6.0 and < 5.0 mg/dL at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, MD, Study Director — Ardea Biosciences, Inc.
Locations (48):
- United States (48):
  - Birmingham, Alabama
  - Gulf Shores, Alabama
  - Mobile, Alabama
  - Glendale, Arizona
  - Peoria, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Gold River, California
  - Irvine, California
  - San Leandro, California
  - San Ramon, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Jacksonville, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Dunwoody, Georgia
  - Honolulu, Hawaii
  - Meridian, Idaho
  - Gurnee, Illinois
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Metairie, Louisiana
  - Jackson, Mississippi
  - Reno, Nevada
  - New York, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Shelby, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Perrysburg, Ohio
  - Willoughby Hills, Ohio
  - Altoona, Pennsylvania
  - Greenville, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Rock Hill, South Carolina
  - Spartanburg, South Carolina
  - Spring Hill, Tennessee
  - Houston, Texas
  - Bountiful, Utah
  - Midlothian, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia